CLINICAL TRIAL: NCT03233958
Title: The Psychosocial Effects of Systemic / Family Constellation: An Observational Follow-up Study
Brief Title: The Psychosocial Effects of Systemic / Family Constellation
Status: Completed | Type: Observational
Sponsor: Károli Gáspár University of the Reformed Church in Hungary (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Principal Investigator, Gergely Sándor Szabó, PhD, Assistant Professor, Károli Gáspár University of the Reformed Church in Hungary
Other Study IDs: 325/2017/P
Record Dates: First submitted 2017-07-25; First posted 2017-07-31 (Actual); Results first posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Mild to Moderate Psychopathological Symptoms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Workshop participants: Participants of systemic / family constellation workshops
  Interventions: Behavioral: Systemic / family constellation

INTERVENTIONS:
Behavioral: Systemic / family constellation — Systemic / family constellation integrates elements from psychodrama, family sculpture, and spontaneous dramatizations of intra- and interpersonal processes, while spatially visualizing family dynamics. Family constellations stimulate change through the following ways: 1) making visible the spatial arrangement of relationships within a conflictual system; 2) providing access to the insights of unrelated third parties regarding the sensations, feelings, and thoughts they experienced while representing family members within the constellation; and 3) making observable (from the outside) and experienceable (from within) the transformation of the problem constellation into the solution constellation [Hunger, Weinhold, Bornhäuser, Link, & Schweitzer, 2015].

SUMMARY:
The purpose of this study is to investigate the psychosocial effects of systemic / family constellation. The method of systemic / family constellation refers to an approach which integrates ideas from family systems therapy with elements from psychodrama. The constellations are conducted in a group based seminar-setting, each seminar lasting two days.

Considering the very limited amount of empirical data on this method, the study design is a simple pre-post one with a 6-months follow-up. The study will be observational: the researchers will not manipulate who receives the intervention; instead they invite all clients (individuals from the general population) attending these therapeutic workshops run independently of the research process. Given the limited amount of evidence on this therapeutic method, special attention will be given to monitor potential adverse outcomes to establish intervention safety.

It is hypothesized that participation in a family constellation seminar might decrease potential psychological symptoms and will not result in adverse outcomes.

DETAILED DESCRIPTION:
Family / systemic constellation therapy is a short-term group psychotherapy aiming to help clients better understand and resolve their conflicts within their personal systems, which in turn might lead to a decrease in psychopathological or functional somatic symptoms. The personal system addressed is most often the family but other inter- or intrapersonal systems (e.g., ego parts, victim-perpetrator dyads) can also be the target of the intervention; the term "family constellation therapy" is used throughout the manuscript in this broader sense. This therapeutic modality was developed in Germany in the early '90s integrating elements of - among others - psychodrama, family sculptures, contextual therapy, and certain South-African aboriginal traditions and has become particularly popular in Europe and South America and even became part of the public health care system in certain countries. Compared to its use by thousands of therapists of various theoretical and professional backgrounds all over the world, little effort has been made to generate empirical data regarding the effectiveness and safety of this intervention.

We believe that the large discrepancy between the relatively high level of penetration into the practice of complementary and alternative medicine versus the low quantity of evidence on effectiveness stems largely from academic psychology's reluctance to engage with at least two metaphysical / anthropological postulates of family constellation therapy. Firstly, the theory of family constellation therapy assumes that an individual's mental and physical health might be significantly influenced by major life events of other members of the personal system even if they lived generations before (e.g., the death of a mother during childbirth might have an effect on her descendants' anxiety level and reproductive success for several generations even if the original event has never been talked about in the descendant's life). While - due to recent developments in epigenetics and the better understanding of transgenerational trauma - this and similar concepts are less shocking to the academic community than they were 3-4 decades ago when family constellation therapy was developed, they are still in sharp contradiction with the common understanding that the etiological factors of any physical or mental illness are to be sought in bio-psycho-social events, situations, or conditions occurring or existing around and after the individual's conception.

The second distinctive feature is that the theory of family constellation therapy assumes that the life-altering, relevant pieces of information are 'stored' and somehow can be 'downloaded' not just automatically and unconsciously by the members of the same system but intentionally by outsiders as well. This accessibility of system-relevant information makes it possible that participants of the single-occasion intervention (who are unknown to each other) are able to perceive and verbalize thoughts, physical perceptions, emotions associated with the history of the system, often unknown even to the recipient of the given constellation. This somewhat 'mystical' re-presentation of unknown facts and hidden dynamics makes it possible for the recipient of the constellation to better understand the etiology of their mental or physical symptoms and intentionally change these very same dynamics. How this storage and access of system-relevant information occurs is highly debated and uncertain; the most-widely held explanation of these processes use the morphic / morphogenic field and -resonance concepts (cf. storage) of the biologist Rupert Sheldrake in combination with the function of mirror neurons (cf. way of accessing stored information by non-members of the system).

Regardless of whether we fully understand the exact mechanisms of action of a therapeutic modality and if its certain assumptions fit the contemporary paradigms of health sciences, we argue that collecting empirical data on an intervention's effectiveness and safety is a public health necessity, especially if it is so widely used as family constellation therapy (and it certainly could provide further impetus to the study of the mechanisms of action and the potential reconsideration of the accuracy of our paradigms).

The very limited number of previous prospective, peer-reviewed studies into family constellation therapy's therapeutic effectiveness reported that the intervention was effective in reducing general, non-diagnosis-specific psychopathology and psychological distress, decreasing the intensity of dermatological symptoms, as well as improving quality of life and functioning in interpersonal relationships. A recent systematic review summarizing both the peer-reviewed and the grey literature on family constellation therapy concluded that further studies into its effectiveness are greatly needed, especially if 1) using at least a mid-term time frame (≥6 months) to evaluate client outcomes, 2) employing active monitoring (not just passive surveillance) of potential iatrogenic effects, and 3) providing information on the presence or absence of therapist effects. The aim of the present study was to collect and analyze further data from the real life setting on family constellation therapy's effectiveness in improving mental health and its tolerability in line with these recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Self-referred and registered for a family constellation workshop with one of the therapists (clinical psychologist / psychiatrist) who were willing to collaborate with the researchers of the present study

Exclusion Criteria:

* Age under 18 years
* Currently suffers from a diagnosed mental disorder
* Participated actively (not merely as a "representative") in a family constellation intervention in the 12 months preceding baseline assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals from the general population who seek help through family constellation seminars for various mild to moderate psychological symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barna Konkoly Thege, PhD, Study Director — Department of Psychiatry, Univeristy of Toronto
Locations (1):
- Károli Gáspár University of the Reformed Church in Hungary, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: Undecided
The investigators have not requested permission from their study participants to make their data available to others to increase participants' sense of confidentiality and so willingness to participate in the study. As a consequence, in case of a data sharing request, the investigators would have to seek for additional explicit permission from the participants. As the investigators have committed to destroy participant contact data after finishing the study, the chances of such data sharing seem slim. However, the investigators are more than happy to conduct alternative analyses based on interested colleagues' suggestions / inquiry and share the raw output (including analytic syntax) of such analyses with those making the inquiry.

REFERENCES:
- [Background] Weinhold J, Hunger C, Bornhauser A, Link L, Rochon J, Wild B, Schweitzer J. Family constellation seminars improve psychological functioning in a general population sample: results of a randomized controlled trial. J Couns Psychol. 2013 Oct;60(4):601-9. doi: 10.1037/a0033539. Epub 2013 Aug 19. PMID 23957767
- [Background] Hunger C, Weinhold J, Bornhauser A, Link L, Schweitzer J. Mid- and long-term effects of family constellation seminars in a general population sample: 8- and 12-month follow-up. Fam Process. 2015 Jun;54(2):344-58. doi: 10.1111/famp.12102. Epub 2014 Sep 29. PMID 25264190
- [Background] Hunger C, Bornhauser A, Link L, Schweitzer J, Weinhold J. Improving experience in personal social systems through family constellation seminars: results of a randomized controlled trial. Fam Process. 2014 Jun;53(2):288-306. doi: 10.1111/famp.12051. Epub 2013 Nov 19. PMID 24251855
- [Background] Konkoly Thege B, Petroll C, Rivas C, Scholtens S. The Effectiveness of Family Constellation Therapy in Improving Mental Health: A Systematic Review. Fam Process. 2021 Jun;60(2):409-423. doi: 10.1111/famp.12636. Epub 2021 Feb 2. PMID 33528854
- [Result] Konkoly Thege B, Somogyi B, Szabo GS. The Effectiveness of Family Constellation Therapy in Reducing Psychopathological Symptoms in a Naturalistic Setting. Psychiatr Danub. 2022 Fall;34(3):497-505. doi: 10.24869/psyd.2022.497. PMID 36256988

RESULTS

PARTICIPANT FLOW:
Groups:
- Family Constellation Participants: Participants of systemic / family constellation workshops
Period: Overall Study
Arm/Group | Family Constellation Participants
Started | 182
Completed | 102
Not Completed | 80

BASELINE CHARACTERISTICS:
Arm/Group | Workshop Participants
Number analyzed (Participants) | 182
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.9 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 152
  Male | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Hungary | 182
General Severity Index of the Brief Symptom Inventory [Mean (Standard Deviation); unit: units on a scale] — The Hungarian version of the Brief Symptom Inventory was used to measure an individual's overall psychopathology level. This tool consists of 53 items covering nine symptom dimensions: somatization, obsessive-compulsive symptoms, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation, and psychoticism. Out of the three global measures of pathology and distress, the General Severity Index (GSI, mean of all items) was used in the present study. The range of this measure is 0-4, higher scores indicating worse mental health (more psychopathological symptoms).
  units on a scale | 0.89 (0.54)

OUTCOME MEASURES:

1. Primary Outcome: Change in General Severity Index Scores on the Brief Symptom Inventory
Description: The Hungarian version of the Brief Symptom Inventory was used to measure an individual's overall psychopathology level. This tool consists of 53 items covering nine symptom dimensions: somatization, obsessive-compulsive symptoms, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation, and psychoticism. Out of the three global measures of pathology and distress, the General Severity Index (GSI, mean of all items) was used in the present study. The range of this measure is 0-4, higher scores indicating worse mental health (more psychopathological symptoms). The range of this measure is 0-4, higher scores indicating worse mental health (more psychopathological symptoms).
Time Frame: Before, 1- and 6-month after the intervention
Population: Participants completing both the baseline and the one- and 6-month follow-up questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Family Constellation Participants
Number analyzed (Participants) | 102
score on a scale
  Baseline | 0.82 (0.51)
  1-month postintervention | 0.56 (0.53)
  6-month postintervention | 0.58 (0.53)
Statistical Analysis 1: Comparison: Family Constellation Participants; Test type: Other — Due to the single group, pre-post design, the analysis simply investigated the effect of time; p < 0.001, ANOVA; Mean Difference (Final Values) = -0.24

2. Secondary Outcome: Change in Scores on the Experience in Personal Social Systems Questionnaire
Description: The Experience in Personal Social Systems Questionnaire assesses social aspects of quality of life (how the respondent feels about their own personal social system). Total score is created by adding all 12 items and the range is 12-72, higher scores indicating better social quality of life.
Time Frame: Before, 1 month after and 6 months after the intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Family Constellation Participants
Number analyzed (Participants) | 102
score on a scale
  Baseline | 44.97 (11.33)
  1-month postintervention | 49.67 (13.76)
  6-month postintervention | 50.52 (13.42)
Statistical Analysis 1: Comparison: Family Constellation Participants; Test type: Other — Due to the single group, pre-post design, the analysis simply investigated the effect of time; p < 0.001, ANOVA; Mean Difference (Final Values) = 5.55

3. Secondary Outcome: Change in Scores on the Patient Health Questionnaire Somatic Symptom Severity Scale (PHQ-15)
Description: The Patient Health Questionnaire Somatic Symptom Severity Scale includes 15 somatic symptoms (headache, stomach pain, chest pain, dizziness, etc.) that account for more than 90% of symptoms seen in primary care (exclusive of upper respiratory symptoms). Total score is the sum of all items, range is 0-30, higher scores indicate more somatic symptoms (worse physical health).
Time Frame: Before, 1 month after and 6 months after the intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Family Constellation Participants
Number analyzed (Participants) | 102
score on a scale
  Baseline | 6.89 (4.26)
  1-month postintervention | 5.55 (4.33)
  6-month postintervention | 6.35 (4.71)
Statistical Analysis 1: Comparison: Family Constellation Participants; Test type: Other — Due to the single group, pre-post design, the analysis simply investigated the effect of time; p = 0.002, ANOVA; Mean Difference (Final Values) = -0.54

4. Secondary Outcome: Change in Scores on the SCOFF Questionnaire
Description: The SCOFF Questionnaire is a brief screener to detect increased risk for eating disorders. The total score is created by summing all five items, leading to a score range of 0-5. Higher scores indicate higher eating disorder risk.
Time Frame: Before, 1 month after and 6 months after the intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Family Constellation Participants
Number analyzed (Participants) | 102
score on a scale
  Baseline | 0.65 (1.00)
  1-month postintervention | 0.55 (0.91)
  6-months postintervention | 0.47 (0.90)
Statistical Analysis 1: Comparison: Family Constellation Participants; Test type: Other — Due to the single group, pre-post design, the analysis simply investigated the effect of time; p = 0.076, ANOVA; Mean Difference (Final Values) = -0.18

5. Secondary Outcome: Change in Scores on ad Hoc Items to Assess Behavioral and Substance-related Addictions
Description: Items assess perceived problem severity with behavioral and substance-related addictions. The total scores is created by summing all four items resulting in a score range of 4-28. Higher scores indicate more severe behavioral and substance-related addiction severity.
Time Frame: Before, 1 month after and 6 months after the intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Family Constellation Participants
Number analyzed (Participants) | 102
score on a scale
  Baseline | 6.73 (3.10)
  1-month postintervention | 6.35 (2.43)
  6-month postintervention | 6.22 (2.65)
Statistical Analysis 1: Comparison: Family Constellation Participants; Test type: Other — Due to the single group, pre-post design, the analysis simply investigated the effect of time; p = 0.147, ANOVA; Mean Difference (Final Values) = -0.51

6. Secondary Outcome: Change in Scores on the Meaning in Life Questionnaire / Presence of Meaning Subscale
Description: The Presence of Meaning Subscale of the Meaning in Life Questionnaire assesses the perceived level of meaning in an individual's life. Total score is created by summing all 5 subscale items resulting a score range of 5-35. Higher scores indicate a higher sense of meaning in life (better mental health).
Time Frame: Before, 1 month after and 6 months after the intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Family Constellation Participants
Number analyzed (Participants) | 102
score on a scale
  Baseline | 22.87 (8.37)
  1-month postintervention | 23.79 (8.95)
  6-month postintervention | 23.94 (8.44)
Statistical Analysis 1: Comparison: Family Constellation Participants; Test type: Other — Due to the single group, pre-post design, the analysis simply investigated the effect of time; p = 0.197, ANOVA; Mean Difference (Final Values) = 1.07

7. Secondary Outcome: Change in Scores on the World Health Organization Wellbeing Index (WBI-5)
Description: The World Health Organization Wellbeing Index captures the general well-being of the individual. Total score is created by summing all 5 items, resulting in a score range of 0-15. Higher scores indicate better overall well-being.
Time Frame: Before, 1 month after and 6 months after the intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Family Constellation Participants
Number analyzed (Participants) | 102
score on a scale
  Baseline | 8.01 (3.27)
  1-month postintervention | 9.10 (3.29)
  6-months postintervention | 9.26 (3.46)
Statistical Analysis 1: Comparison: Family Constellation Participants; Test type: Other — Due to the single group, pre-post design, the analysis simply investigated the effect of time; p < 0.001, ANOVA; Mean Difference (Final Values) = 1.25

8. Secondary Outcome: Participant-perceived Iatrogenic Effects
Description: Qualitative responses on the perceived iatrogenic effects of the intervention were collected using-open ended, ad hoc questions.
Time Frame: 1 month after and 6 months after the intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Workshop Participants
Number analyzed (Participants) | 102
Participants
  1 month | 11
  6 months | 17

ADVERSE EVENTS:
Time Frame: 6 months postintervention
Description: Two items were developed by the investigators to screen for adverse outcomes: "Have you experienced any negative change in relation to your mental or physical health during or since the family constellation workshop?". If respondents answered affirmatively, it was also asked if they believed the changes were associated with the intervention (yes/no/unsure). Below we report all adverse events, including those participants were sure were not related to the intervention.
Arm/Group | Workshop Participants
All-Cause Mortality (participants affected / at risk) | 0/102
Serious Adverse Events (participants affected / at risk) | 0/102
Other Adverse Events (participants affected / at risk) | 17/102
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Workshop Participants (N=102)
Negative mental health outcomes (Psychiatric disorders) | 7 (7) — E.g., slightly more addictive symptoms, increased tensions in marriage, increased fear of aging
Negative physical health outcomes (Endocrine disorders) | 8 (8) — E.g., unintended weight gain, exhaustion, or hypothyroidism
Combined mental and physical negative outcomes (Psychiatric disorders) | 2 (2) — Avolition combined with exhaustion, increased negative affect in combination with unintended weight gain and exhaustion

LIMITATIONS AND CAVEATS:
The most important shortcoming of the present study is the non-controlled nature of its design and thus the possibility that the reported beneficial changes are the results of external factors. A further limitation of the present study is the low participation rate of men (even if it corresponds to anecdotic evidence on the real-life gender ratio of participants) and the large attrition rate limiting the generalizability of the findings to all family constellation participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-06-19): https://cdn.clinicaltrials.gov/large-docs/58/NCT03233958/Prot_SAP_ICF_000.pdf